CLINICAL TRIAL: NCT06558331
Title: Comparison of the Effects of ESP Block and Paravertebral Block on the Quality of Postoperative Recovery (QoR-15T) in Patients Undergoing Video-Assisted Thoracoscopic Surgery (VATS)
Brief Title: Quality of Postoperative Recovery (QoR-15T) in Patients Undergoing Video-Assisted Thoracoscopic Surgery (VATS)
Status: Recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Cansu KILINC BERKTAS, Specialist MD, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2024-245
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-08

CONDITIONS: Video-Assisted Thoracic Surgery
Keywords: Video-Assisted Thoracic Surgery; perioperative care; patient-reported outcome measures; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESP Group: After the patients are taken to the operating table and the necessary ASA monitoring is performed, erector spinae plane block (ESP) is performed on the side where surgery will be performed from the T4-T5 thoracic vertebrae level for peroperative analgesia with ultrasound (USG), depending on the clinician's experience and the USG image.
  Interventions: Other: Preoperative Quality of Recovery-15 (QoR-15T); Other: Postoperative 24th hour Quality of Recovery-15 (QoR-15T)
- Paravertebral Group: After the patients are taken to the operating table and the necessary ASA monitoring is performed, paravertebral block is performed on the side where surgery will be performed from the T4-T5 thoracic vertebrae level for peroperative analgesia with ultrasound (USG), depending on the clinician's experience and the USG image.
  Interventions: Other: Preoperative Quality of Recovery-15 (QoR-15T); Other: Postoperative 24th hour Quality of Recovery-15 (QoR-15T)

INTERVENTIONS:
Other: Preoperative Quality of Recovery-15 (QoR-15T) — The quality of recovery score (QoR)-15 questionnaire, preoperative
Other: Postoperative 24th hour Quality of Recovery-15 (QoR-15T) — The quality of recovery score (QoR)-15 questionnaire, postoperative 24th hour

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive technique that provides faster recovery after thoracic surgery. Techniques such as thoracic paravertebral block, Erector Spina Plane Expansion (ESP block) are accepted as loco-regional techniques for VATS. The quality of recovery after anesthesia (QoR) is an important information of the early health components of patients after surgery. QoR-15 offers a valid, reliable, sensitive and easy-to-use method for recovery after surgery. We aimed to investigate the relationship between QoR-15 score and postoperative pain temperature after Video-Assisted Thoracoscopic Surgery (VATS) ESP block and paravertebral spread.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive technique that provides faster recovery after thoracic surgery. Techniques such as thoracic paravertebral block, Erector Spina Plane Expansion (ESP block) are accepted as loco-regional techniques for VATS. Despite the improvement in invasiveness against thoracotomy treatment, postoperative pain after VATS was still moderate to severe. In order to accelerate the recovery of patients, a multimodal analgesic should be carefully planned and where it will be beneficial. The quality of recovery after anesthesia (QoR) is an important information of the early health components of patients after surgery. The performance of QoR-15 has been translated into Turkish and validation studies have been conducted on its products. QoR-15 offers a valid, reliable, sensitive and easy-to-use method for recovery after surgery. We aimed to investigate the relationship between QoR-15 score and postoperative pain temperature after Video-Assisted Thoracoscopic Surgery (VATS) ESP block and paravertebral spread.

ELIGIBILITY:
Inclusion Criteria:

* ASA1-3
* Patient undergoing Video Assisted Thoracoscopic Surgery (VATS)
* Over 18 years of age

Exclusion Criteria:

* Sympathectomy, lobectomy and pneumonectomy surgery using Video Assisted Thoracoscopic Surgery (VATS)
* Cases that started with Video Assisted Thoracoscopic Surgery (VATS) but were converted to thoracotomy,
* Patients who were uncooperative,
* Patients who refused to participate in the study,
* Presence of a neuropsychiatric disorder that could bias QoR-15T measurements or emergency surgical intervention,
* Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Over 18 years of age
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
Effect of ESP block and paravertebral block on QoR-15 Quality of Recovery in VATS surgery | 24 hour
  To demonstrate the effect of ESP block and paravertebral block on patient recovery at 24 hours using the Quality of Recovery-15 (QoR-15) scale in patients undergoing Video-Assisted Thoracoscopic Surgery (VATS), Complication,
Pain score with Numeric Rating Scale (NRS score), | 1 day
  The NRS is a one-dimensional scale using 11 numbers (0 to 10) to measure pain intensity. The patient is asked to choose the number that best reflects the pain intensity, with 0 = no pain and 10 = the worst (unbearable) pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam Ve Sakura Şehir Hastanesi, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol